CLINICAL TRIAL: NCT00908973
Title: Gut Hormone Response, Appetite and Intestinal Transit Time in Good and Poor Weight Responders 1-2 Years After Gastric Bypass
Brief Title: Gut Hormone Response, Appetite and Intestinal Transit Time in Good and Poor Weight Responders After Gastric Bypass
Acronym: RnonR
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Carsten Dirksen, MD PhD student, Hvidovre University Hospital
Other Study IDs: RnonR
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
Keywords: Obesity; Gastric bypass; Gut hormone; Intestinal transit time
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum specimens are retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Good responders: Excess weight loss of > 60% 1 year after gastric bypass surgery
- Poor responders: Excess weight loss of =< 50% 1 year after gastric bypass surgery
- Lean controls: Non-gastric bypass operated lean individuals, matched for age and sex

SUMMARY:
The aim of the study is to describe differences in meal-stimulated gut hormone response, appetite and intestinal transit time between good and poor responders 1-2 years after Gastric Bypass surgery for obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* Completed laparoscopic gastric bypass surgery without complications (cases)
* No previous gastric bypass surgery (controls)

Exclusion Criteria:

* Diabetes
* Disease or treatment interfering with appetite or gastrointestinal motility
* Pregnancy or breastfeeding
* Excess weight loss 1 year after gastric bypass > 50% and =< 60% (cases)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Case subjects are recruited from the outpatient clinic of endocrinology at Hvidovre University Hospital. Control subjects are recruited through announcement in local newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, MD, Principal Investigator — Dept. of Endocrinology, Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark
Locations (1):
- Department of Endocrinology at Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark